CLINICAL TRIAL: NCT05255120
Title: The Effect of Systematic Preoperative Preparation on the Outcome of Benign Hysterectomy: a Prospective Intervention Study
Brief Title: Hysterectomy - A Regional Intervention Study
Acronym: HYSTERI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Preben Kjolhede, MD, professor, Professor, University Hospital, Linkoeping
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYSTERI
Record Dates: First submitted 2022-02-04; First posted 2022-02-24 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Benign Hysterectomy; Postoperative Recovery; Preoperative Planning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensified preoperative information (Experimental): The patient participating in the intervention group is evaluated preoperatively based on an algorithm. This information is designed according to a checklist which includes how the procedure is performed, rules of conduct in connection with and after the procedure and what the patient can expect after surgery.
  Interventions: Other: Intiensified structured perioperative information
- Control group (No Intervention): The patient who participates in the control group receives information about participation in the study as a control, ie without information about the intervention. The patient will then be planned for the procedure according to current, local routines.

INTERVENTIONS:
Other: Intiensified structured perioperative information — The doctor takes a medical history and examines the patient according to regular routines, but uses the algorithm as support in deciding on the surgical method. After the doctor's visit, the patient must see a research nurse to receive the intensified preoperative information about hysterectomy. This information is designed according to a checklist. The patient can also download a mobile application. The study-specific mobile application (app) contains information about hysterectomy. The information is structured in three parts - Before the Operation, At the Hospital and After the Operation. A timeline describes the activities and events that occur before, around and after the operation. Within each section there are several information links, with eg checklists.
  Arms: Intensified preoperative information

SUMMARY:
Approximately 4,000 procedures with hysterectomy for benign indication are performed annually in Sweden. There are large differences in preoperative information, planning of surgery and surgical technique. A structured approach including the use of mobile phone technology can possibly improve patient information and patient involvement. Our purpose is to to evaluate whether systematic preoperative preparation improves the outcome of elective hysterectomy on benign indication.

DETAILED DESCRIPTION:
Background Approximately 4,000 procedures with hysterectomy for benign indication are performed annually in Sweden. There are large differences between clinics in Sweden in the proportion of hysterectomies conducted using minimally invasive surgery. There is no uniformity in the planning of surgery. Patient-reported outcome measures, such as satisfaction and postoperatively unexpected symptoms, are important in assessing the outcome of surgery. Patient-reported measurements are, besides other factors, dependent on preoperative information. Mobile phone technology can possibly improve patient information and patient involvement.

Purpose

To evaluate whether a systematic preoperative preparation improves the outcome of elective hysterectomy on benign indication. The work consists of three parts with the following purposes:

Sub-study 1: To evaluate the effect of a preoperative algorithm for determining the most appropriate method of hysterectomy on the proportion undergoing surgery as a minimally invasive procedure and on the frequency of complications.

Sub-study 2: To compare patient-reported outcome measures, including unexpected symptoms, recovery, and satisfaction, in women who receive systematic preoperative information from specially trained staff and a mobile application with targeted education on the procedure, with women who receive information according to normal routines.

Sub-study 3: To investigate how women experience digitized information via a mobile application in connection with surgery.

Participating centers Departments of obstetrics and gynecology at the hospitals in Norrköping, Jönköping, Eksjö, Värnamo, Västervik, Kalmar and Växjö.

Schedule The study starts in September 2020. Recruitment of patients is planned to take two years.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 - 55 years old.
* Women undergoing hysterectomy for benign indication.
* Women with ASA 1 - 3.
* Women who understand and can express themselves in Swedish.
* Women who, by signing "Informed Consent", agree to participate in the study after written and oral information.
* Women who participate and respond to the surveys in the GynOp register.
* Women who have access to an I-phone, smartphone, computer or tablet and who can use the study-specific mobile application. (Does not apply to sub-study 1).

Exclusion criteria

* Women where both ovaries are removed during the operation.
* Women undergoing hysterectomy for prolapse indication.
* Women undergoing hysterectomy for cancer prophylactic indication.
* Women undergoing hysterectomy for gender reassignment purposes.
* Women with intellectual disabilities to such an extent that they can not fill in the relevant questionnaires etc. or if they do not understand the meaning of participating in the study or where there may be ethical doubts about the patient's participation in the study.
* Women who have a mental illness of such severity that the doctor in charge considers it inappropriate for the patient to be included in the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients undergoing hysterectomy
Enrollment: 230 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Unexpected postoperative symtoms | Up to one year postoperatively
  Proportion of patients with unexpected symptoms.
Proportion minimally invasive hysterectomy | Retrospecive data 5 years before study start until completion of prospective study
  Proportion of women undergoing hysterectomy as a minimally invasive procedure

SECONDARY OUTCOMES:
Complication | Up to one year postoperatively
  Numbers of and types of patient reported complications
Lenght of stay | Day of surgery until discharge from hospital pre- and during the intervention
  Hospital length of stay in connection with surgery
Sick leave | Day of discharge from hospital after surgery until return to normal work, maximal one year
  return to work measured as actual sick leave length
Recovery | Day of surgery until normal ADL, maximal one year
  time to normal daily activity (ADL)
Health related quality of life | Preoperatively up to one year postoperatively
  Measured with EuroQol EQ-5D-3L health index comprising of two parts. Part A Scale -0.5941 to 1. A higher number indicates better quality of life. Part B. EuroQol visual analoque scale EQ-VAS. Scale 0-100. A higher number indicates better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kjölhede, MD PhD, Study Chair — University Hospital, Linköing; Lollo Makdessi, MD, Study Chair — Vrinnevi Hospital, Norrköping
Locations (2):
- Sweden (2):
  - University Hospital, Linköping
  - Vrinnevisjukhuset, Norrköping

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorkstrom LM, Wodlin NB, Nilsson L, Kjolhede P. The Impact of Preoperative Assessment and Planning on the Outcome of Benign Hysterectomy - a Systematic Review. Geburtshilfe Frauenheilkd. 2021 Feb;81(2):200-213. doi: 10.1055/a-1263-0811. Epub 2021 Feb 8. PMID 33574624